CLINICAL TRIAL: NCT05258565
Title: Tissue Plasminogen Activator (tPA) Therapy for Acute Ischemic Stroke in Covid -19 and Non Covid -19 Patients
Brief Title: TPA in Acute Stroke With COVID Verus Non-COVID-19 Patients
Acronym: rTPA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, clinical professor, Assiut University
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: TPA in acute stroke
Record Dates: First submitted 2022-02-21; First posted 2022-02-28 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acute ischemic stroke without covid -19 infection (Active Comparator): Administration of IV tPA: the dose of activase is ,9 mg /kg (not exceeding 90 mg total treatment dose) Infused over 90 minutes.
  Interventions: Drug: IV tPA (Activase)
- acute ischemic stroke associated with covid -19 infection (Active Comparator): Administration of IV tPA: the dose of activase is, 9 mg /kg (not exceeding 90 mg total treatment dose) Infused over 90 minutes.
  Interventions: Drug: IV tPA (Activase)

INTERVENTIONS:
Drug: IV tPA (Activase) — Any patients eligible came with acute ischemic stroke with or without COVID-19 infection within the time window for thrombolytic therapy (within 4 hours of onset)
  Other Names: IV tissue plasminogen activator

SUMMARY:
The investigator will recruit consecutively all patients coming with acute ischemic stroke either with or without COVID -19 infection and suitable for IV injection with Tissue plasminogen activators according to guideline and inclusion criteria of tPA.

Aswan University Hospital.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS) is a time sensitive medical emergency and a leading cause of morbidity and mortality worldwide. Intravenous (IV) recombinant tissue plasminogen activator (IV alteplase) is currently the only proven effective medication for the treatment of AIS with promising adjuvant medications currently under investigation.(Gottula et al, 2021).

Intravenous tissue plasminogen activator (tPA) is used to treat acute stroke because of its thrombolytic activity and its ability to restore circulation to the brain. (Wang, et. al, 1998). However tPA administration, especially delayed administration is associated with increased intracranial hemorrhage, hemorrhagic transformation and mortality. (Jong, 2019) Acute cerebrovascular disease, particularly ischemic stroke, has emerged as a serious complication of infection by the severe acute respiratory syndrome coronavirus that caused by the Coronavirus disease-2019 (COVID-19). Such specificities include a propensity towards large vessel occlusion, multi-territory stroke, and involvement of otherwise uncommonly affected vessels. The pathogenesis and optimal management of ischemic stroke associated with COVID-19 still remain uncertain, but emerging evidence suggest that cytokine storm-triggered coagulopathy and endotheliopathy represent possible targetable mechanisms. (Vogrig, et. al, 2021).

Anew study was done in United States in 2020, included 13 patients presented with acute ischemic stroke and systemic symptoms consistent with covid-19 were treated with IV tPA. 61.5% of patients improved at follow up, Neither of them complicated with systemic or symptomatic intracranial hemorrhages.(Carneiro, et. al, 2020). IV tPA may be safe and efficacious in COVID -19 but larger studies are needed to validate these results (Carneiro, et. al, 2020).

The purpose of this study is to compare between the safety and efficacy of tPA management of ischemic stroke in Covid-19 and non covid-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as acute ischemic stroke NIHSS<25
* Symptoms onset less than 4.5 hours (3hours in diabetic or having a previous stroke) before beginning treatment.

Exclusion Criteria:

* History of:

  * A previous ischemic stroke or severe head trauma in previous 3 months.
  * Previous intracranial hemorrhage .
  * Intracranial neoplasm or gastrointestinal malignancy.
  * Gastrointestinal hemorrhage in previous 3weeks.
  * Intracranial or intra spinal surgery in previous 3months

Clinically:

* Symptoms suggestive of subarachnoid hemorrhage.
* Persistent blood pressure elevation, systolic > 185 or diastolic >110 mmHg.
* Active internal bleeding.
* Presentations consistent with infective endocarditis.
* Stroke known or suspected to be associated with aortic arch dissection.
* Acute bleeding diathesis, including but not limited to conditions defined under hematologic.

Hematologic:

* Platelet count <100.000 \ mm3
* Current anticoagulant use with INR>1.7 or PT>15sec or PTT> 40sec.
* Therapeutic doses of low molecular weight received in 24 hours (not include the prophylactic doses).

Head CT:

* Evidence of hemorrhage.
* Extensive regions of obvious hypo density

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
primary out come | 2 months
  Barthel Index scale BIS (pre-post drug administration and 2 month later)The Barthel includes 10 personal activities: feeding, personal toileting, bathing, dressing and undressing, getting on and off a toilet, controlling bladder, controlling bowel, moving from wheelchair to bed and returning, walking on level surface (or propelling a wheelchair if unable to walk) and ascending and descending stairs.
  The original Index is a three-item ordinal rating scale completed by a therapist or other observer in 2-5 minutes. Each item is rated in terms of whether the patient can perform the task independently, with some assistance, or is dependent on help based on observation (0=unable, 1=needs help, 2=independent). The final score is x 5 to get a number on a 100 point score. Proposed guidelines for interpreting Barthel scores are that scores of 0-20 indicate "total" dependency, 21-60 indicate "severe" dependency, 61-90 indicate "moderate" dependency, and 91-99 indicates "slight" dependency.

SECONDARY OUTCOMES:
secondary outcome | 2 months
  NIHSS (pre-post drug administration and 2 month later a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items( Level of Consciousness ,Horizontal Eye Movement, Visual field test, Facial Palsy, Motor Arm, Motor Leg, Limb Ataxia ,Sensory, Language and Speech)
  , each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.Score 0 means No stroke symptoms. score 1-4 means Minor stroke .Score 5-15 means Moderate stroke. score 16-20 means Moderate to severe stroke. Score 21-42 means Severe stroke

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Aswan University Hospital, Aswān
  - Assiut University Hospital, Asyut

REFERENCES:
- See also: • Gottula AL, Barreto AD, Adeoye O. Alteplase and Adjuvant Therapies for Acute Ischemic Stroke. Semin Neurol. 2021 Feb;41(1):16-27. doi: 10.1055/s-0040-1722720. Epub 2021 Jan 20. PMID: 33472270.. — https://pubmed.ncbi.nlm.nih.gov/33472270/
- See also: • Wang YF, Tsirka SE, Strickland S, Stieg PE, Soriano SG, Lipton SA.Tissue plasminogen activator (tPA) increases neuronal damage after focal cerebral ischemia in wild-type and tPA-deficient mice. — https://pubmed.ncbi.nlm.nih.gov/9461198/
- See also: • Vogrig A, Gigli GL, Bnà C, Morassi M. Stroke in patients with COVID-19: Clinical and neuroimaging characteristics. Neurosci Lett. 2021 Jan 19;743:135564. doi: 10.1016/j.neulet.2020.135564. Epub 2020 Dec 19. PMID: 33352277; PMCID: PMC7749733. — https://pubmed.ncbi.nlm.nih.gov/33352277/
- See also: • Kim, Jong S. "tPA Helpers in the Treatment of Acute Ischemic Stroke: Are They Ready for Clinical Use?." Journal of stroke vol. 21,2 (2019): 160-174. doi:10.5853/jos.2019.00584 — https://pubmed.ncbi.nlm.nih.gov/31161761/
- See also: Intravenous tPA for Acute Ischemic Stroke in Patients with COVID-19. J Stroke Cerebrovasc Dis. 2020 Nov;29(11):105201. doi: 10.1016/j.jstrokecerebrovasdis.2020.105201. Epub 2020 Jul 27. PMID: 33066885; PMCID: PMC7383145. — https://scholarlycommons.henryford.com/neurology_articles/478